CLINICAL TRIAL: NCT02517359
Title: A Randomized, Double Blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Treatment With Single and Repeat Doses of Inhaled RV6153 in Healthy Subjects and Subjects With Stable Asthma.
Brief Title: A Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Repeat Doses of RV6153
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Preset pharmacokinetic stopping criteria met at lower doses than expected.
Sponsor: Respivert Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SFT001; 2015-000440-41 (EudraCT Number)
Record Dates: First submitted 2015-07-28; First posted 2015-08-07 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Asthma; Healthy Volunteers
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Single dose, healthy volunteers (Experimental)
  Interventions: Drug: RV6153 single dose; Drug: RV6153 matching placebo single dose
- 14 day repeat dose, healthy volunteers (Experimental)
  Interventions: Drug: RV6153 14 day repeat dose; Drug: RV6153 matching placebo 14 day repeat dose
- 28 day repeat dose, healthy volunteers (Experimental)
  Interventions: Drug: RV6153 28 day repeat dose; Drug: RV6153 matching placebo 28 day repeat dose
- 14 day repeat dose, asthma patients (Experimental)
  Interventions: Drug: RV6153 14 day repeat dose; Drug: RV6153 matching placebo 14 day repeat dose
- 14 day repeat dose, smokers (Experimental)
  Interventions: Drug: RV6153 14 day repeat dose; Drug: RV6153 matching placebo 14 day repeat dose

INTERVENTIONS:
Drug: RV6153 single dose — Safety and tolerability of single doses
  Arms: Single dose, healthy volunteers
Drug: RV6153 matching placebo single dose — Safety and tolerability of single doses
  Arms: Single dose, healthy volunteers
Drug: RV6153 14 day repeat dose — Safety and tolerability of repeat doses
  Arms: 14 day repeat dose, asthma patients; 14 day repeat dose, healthy volunteers; 14 day repeat dose, smokers
Drug: RV6153 matching placebo 14 day repeat dose — Safety and tolerability of repeat doses
  Arms: 14 day repeat dose, asthma patients; 14 day repeat dose, healthy volunteers; 14 day repeat dose, smokers
Drug: RV6153 28 day repeat dose — Safety and tolerability of repeat doses
  Arms: 28 day repeat dose, healthy volunteers
Drug: RV6153 matching placebo 28 day repeat dose — Safety and tolerability of repeat doses
  Arms: 28 day repeat dose, healthy volunteers

SUMMARY:
RV6153 is a new medicine being developed for possible treatment of asthma and smoking related lung disease (also known as chronic obstructive pulmonary disease - COPD).

The main purpose of this study is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and repeat doses of RV6153

ELIGIBILITY:
Inclusion Criteria:

Cohorts 1 to 13 (all subjects)

* Subject must be a man or woman aged between 18 to 65 years of age, inclusive: Women of non-childbearing potential only - defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile or permanently sterilised. Men who are willing and able to use suitable contraception methods listed in Section 4.5.1, from the time of the first dose of study medication until 90 days after discharge from the study.
* A woman must have a negative serum β human chorionic gonadotropin (β-hCG) test at screening and a negative urine pregnancy test at Day -1.
* Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Each subject must sign an informed consent form (ICF)
* Body weight ≥50 kg and BMI within the range 19-29 kg/m2 (inclusive).
* Average QTcF <450 msec at screening and Day -1 visits
* Vital sign assessments within normal ranges.

Cohorts 1 to 11 and 13 (healthy volunteers and smokers only)

* Healthy as determined by a physician, based on a full medical evaluation including medical history, physical examination, laboratory tests.
* Spirometry readings (FEV1 and FVC) to be ≥80% predicted value and FEV1/FVC ratio >0.7 at screening.

Cohort 12 (asthma patients only)

* Documented history of asthma, first diagnosed at least 6 months prior to the screening visit.
* Currently being treated with daily standard of care asthma therapy
* Have a diagnosis of asthma confirmed at screening by bronchodilator reversibility.
* Have stable asthma based on physician assessment at screening and prior to randomisation, with no asthma exacerbation requiring augmentation of therapy in the 12 weeks prior to screening and no hospitalization or visit to accident and emergency for asthma in the 12 months prior to screening.
* Have a pre-bronchodilator forced expiratory volume in the first second (FEV1) ≥60% and ≤85% of predicted normal value at screening.
* Subject must be otherwise healthy on the basis of full medical evaluation performed at screening.

Cohort 13 (smokers only)

* Subjects who are current daily cigarette smokers.

Exclusion Criteria:

Cohorts 1 to 13 (all subjects)

* Upper or lower respiratory tract infection within 4 weeks of the screening visit and prior to randomisation.
* A positive pre-study hepatitis B surface antigen or positive hepatitis C antibody result at screening.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities.
* Positive test for alcohol or drugs of abuse.
* Use of prescription medications within 14 days prior to the screening visit and agree not to use prescription medications throughout the duration of the study.
* Are taking over the counter (OTC) medications for 14 days prior to Screening visit and agree to refrain from taking such medications throughout the study.
* History of regular alcohol consumption within 6 months of the study
* Definite or suspected history of drug or alcohol abuse within the previous 5 years.
* A positive test for HIV antibody.
* Received an experimental drug or used an experimental medical device within 3 months or within a period less than five times the drug's half-life before the first dose of the study drug is scheduled.
* Allergy to any of the active or inactive ingredients (including lactose and milk protein intolerance) in the study medication.
* History of drug, or other allergy that would contraindicate their participation.
* A disclosed history or one known to the Investigator, of significant non-compliance in previous investigational studies or with prescribed medications.
* Donated blood or blood products or had substantial loss of blood (more than 500 mL) within 3 months before the first administration of study drug or intention to donate blood or blood products during the study.
* Subject is mentally or legally incapacitated.
* Subject is an employee of the Sponsor or contract research organization (CRO), or a relative of an employee of the Sponsor or CRO.
* Unable or unwilling to undergo multiple venipuncture procedures or the subject has poor access to veins suitable for cannulation.
* Any other reason that the Investigator considers makes the subject unsuitable to participate.

Cohorts 1 to 11 (healthy subjects only)

* Any acute or chronic illness or clinically relevant abnormality identified on the screening medical assessment.
* The subject is a smoker or has smoked or used nicotine-containing products (including e-cigarettes or other nicotine containing products) within the 6 months prior to screening or has a smoking history of ≥5 pack years.
* Positive urine cotinine test at the screening visit indicative of smoking or use of tobacco or nicotine-containing products.

Cohort 12 (asthma patients only)

* Has ever had an episode of life-threatening asthma defined as respiratory arrest, intubation for asthma, or ICU admission for asthma
* Has been hospitalized for greater than 24 hours due to asthma in the 5 years prior to the study.
* Has experienced an asthma exacerbation in the 3 months prior to screening (and prior to randomisation) requiring management with systemic or injectable steroids.
* Has uncontrolled (severe) asthma and/or use of the study prohibited asthma medications.
* The subject is a smoker (regular or irregular), or has smoked or used nicotine-containing products (including e-cigarettes) within the 6 months prior to screening (or a smoking history ≥10 pack years).
* Positive urine cotinine test at the screening visit, and at Day -1, indicative of smoking or use of tobacco or nicotine-containing products.

Cohort 13 (smokers only)

* Any acute or chronic illness, including a diagnosis of COPD, or clinically relevant abnormality identified on the screening medical assessment.
* Subjects who are unable to produce a viable sputum sample at screening
* Subjects whose primary consumption of tobacco is via methods other than cigarettes. Primary methods of tobacco consumption that are excluded include, but are not limited to pipes, cigars and e-cigarettes.
* Urinary cotinine levels at screening <30 nanograms (ng)/mL.
* Subjects who have asthma or a history of asthma (except in childhood and which has now remitted).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-07; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of single and repeat doses assessed by incidence of treatment emergent adverse events | Up to 29 days post final dose
  Assessment of the number of adverse events reported by subjects following dosing
Safety and tolerability of single and repeat doses assessed by ECG (12-lead ECG) | Up to 29 days post final dose
  12-lead ECGs will be obtained using an ECG machine that automatically calculates heart rate and measures PR, QRS, QT, and QTcB/QTcF intervals. ECGs will be measured after resting for 5 minutes
Safety and tolerability of single and repeat doses assessed by vital sign measurement (blood pressure & heart rate) | Up to 29 days post final dose
  Blood pressure heart rate will be assessed together using an automated device after resting for 5 minutes. Blood pressure will include systolic and diastolic measurements.
Safety and tolerability of single and repeat doses assessed by respiration rate | Up to 29 days post final dose
  Respiration rate will be measured after resting for 5 minutes
Safety and tolerability of single and repeat doses assessed by temperature | Up to 29 days post final dose
  Temperature will be measured orally
Safety and tolerability of single and repeat doses assessed by spirometry | Up to 29 days post final dose
  Pulmonary function test measured from forced expiratory volume in 1 second (FEV1). Pulmonary function test will be repeated until three technically acceptable measurements have been made.
Safety and tolerability of single and repeat doses by assessment of clinical laboratory tests | Up to 29 days post final dose
  Clinical laboratory tests include haematology, clinical chemistry, urinalysis and additional parameters
Pharmacodynamic (PD) effect of repeat doses of RV6153 assessed by sputum cell biomarkers | Cohort 13 (subjects who smoke) only - assessments at screening and Days 1, 7 & 14
  Sputum samples will be collected to evaluate PD effects of repeat doses of RV6153 by assessment of phosphatidylinositol biphosphate (PIP2) and phosphatidylinositol triphosphate (PIP3).

SECONDARY OUTCOMES:
Plasma RV6153 levels | Cohorts 1-9: Day 1, 10 samples, Days 2,8,15&29, 1 sample per day; Cohorts 10, 12 & 13: Days 1,7&14, 10 samples per day, Days 2,8-13,1,21,28&42, 1 sample per day; Cohort 11: Days 1,14&28, 10 samples per day, Days 7,21,26,27,29,35,42&56, 1 sample per day

OTHER OUTCOMES:
Sputum markers of inflammation | Cohort 13 (subjects who smoke) only - assessments at screening and Days 1, 7 & 14
  Sputum samples will be collected to evaluate effects on inflammation by assessment of myeloperoxidase, IL-6, IL-8, TNF alpha and other exploratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Christopher O'Brien, MD, PhD, FCCP, Study Director — Sponsor GmbH
Locations (2):
- United Kingdom (2):
  - Manchester
  - Nottingham